CLINICAL TRIAL: NCT04041882
Title: 68Ga-DOTATATE PET/CT for Detection and Evaluation of Neuroendocrine Tumor
Brief Title: 68Ga-DOTATATE PET/CT in Neuroendocrine Tumor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM022
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATATE PET/CT (Experimental): Inject 68Ga-DOTATATE and then perform PET/CT scan
  Interventions: Drug: 68Ga-DOTATATE

INTERVENTIONS:
Drug: 68Ga-DOTATATE — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-DOTATATE. Tracer doses of 68Ga-DOTATATE will be used to image lesions of NET PET/CT scan.

SUMMARY:
Somatostatin receptor(SSTR) was expressed in neuroendocrine tumor cells and SSTR-targeting molecular imaging(68Ga-DOTATATE PET/CT) could be a promising technique to evaluate the primary tumor and metastatic lesions of neuroendocrine tumors with higher accuracy. This prospective study is going to investigate whether radiolabeled somatostatin analogs 68Ga-DOTATATE PET/CT may be valuable for diagnosis, risk stratification, and prognostic evaluation of neuroendocrine tumors and compared it with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Neuroendocrine tumor(NET)can be derived from endocrine glands, endocrine tissues and endocrine cells from any parts of body. Due to its occult onset and heterogeneity, it is hard to be detected by conventional imaging like CT and it is often at late stage when diagnosed. New imaging modality such as 18F-FDG PET/CT have been well-accepted as a practical way to evaluate the aggressive of tumor. 18F-FDG PET/CT has been used to improve the efficacy in assessing the extent and severity of NET, but the diagnostic accuracy of 18F-FDG PET/CT decreased in low proliferation tumor cells and inflammation. Recent studies showed somatostatin receptor (SSTR) was expressed in NET cells and SSTR-targeting molecular imaging-68Ga-DOTATATE PET/CT could be a promising technique to evaluate the extent of NET with higher accuracy. Especially in some well differentiated tumor, 18F-FDG PET/CT can be negative, while 68Ga-DOTATATE PET/CT can be positive. However, the results can be varied in these two imaging modalities and characterized this disease at multiple levels such as clinical presentation, biologic characteristics, treatment response, and clinical outcome.This prospective study is going to investigate whether 68Ga-DOTATATE PET/CT may be superior to 18F-FDG PET/CT for diagnosis, risk stratification, and prognostic evaluation of NET.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated NET patients previously performed 18F-FDG PET/CT signed written consent.

Exclusion Criteria:

* pregnancy breastfeeding known allergy against TATE any medical condition that in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 3 years
  SUVmax of focal lesions are measured on 68Ga-DOTATATE PET/CT. The SUVmax higher than that of the normal liver tissue is defined as positive.
Diagnostic value | through study completion, an average of 3 years
  Diagnostic value of 68Ga-DOTATE PET/CT for NET in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Diagnostic value in different grades/types of NET | through study completion, an average of 3 years
  Diagnostic value of 68Ga-DOTATATE PET/CT in ectopic ACTH-secreting tumor, insulinoma, glucagonoma and so on.
Overall Survival(OS) | 1 year and 5 years after been diagnosed
  Analysis of OS for patients receiving 68Ga-DOTATATE PET/CT
Progressive free survival(PFS) | 1 year and 5 years after been diagnosed
  Analysis of PFS for patients receiving 68Ga-DOTATATE PET/CT
SSTR expression/Ki67 and SUV | through study completion, an average of 3 years
  Correlation between SSTR expression/Ki 67 and SUV in PET
Risk stratification | through study completion, an average of 3 years
  Analysis of risk factors and OS/PFS

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PhD, Study Chair — Peking Union Medical College Hopital, Chinese Academy of Medical Science
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Zang J, Yang Y, Ling Q, Wu H, Wang P, Lu L, Zhu Z. Head-to-head comparison of 68Ga-DOTATATE PET/CT and 18F-FDG PET/CT in localizing tumors with ectopic adrenocorticotropic hormone secretion: a prospective study. Eur J Nucl Med Mol Imaging. 2021 Dec;48(13):4386-4395. doi: 10.1007/s00259-021-05370-8. Epub 2021 Jun 19. PMID 34146130